CLINICAL TRIAL: NCT06707311
Title: A Comparative Study of Different Traditional and Bioactive Indirect Pulp Capping Materials on Dentin Hypersensitivity.In-vivo Study
Brief Title: A Comparative Study of Different Traditional and Bioactive Indirect Pulp Capping Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Badr University (Other)
Responsible Party: Principal Investigator, Mai Salah Ibrahim Afifi Elgohary, Lecturer in BADR University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUC-IACUC-240623-102
Record Dates: First submitted 2024-11-21; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Deep Carious Lesions; Caries Class I; Caries Class II

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- patients received calcium hydroxide with resin composite (Active Comparator): patients received calcium hydroxide lining material then restored with resin composite
  Interventions: Other: patients received calcium hydroxide with glass ionomer restorative material
- patients received TheraCal LC with resin composite (Active Comparator): patients received TheraCal LC lining material then restored with resin composite
  Interventions: Other: patients received TheraCal LC with glass ionomer restorative material
- patients received universal bonding with resin composite (Active Comparator): patients received universal bonding as lining material then restored with resin composite
  Interventions: Other: patients received universal bonding with glass ionomer restorative material
- patients received bioactive bonding with resin composite (Active Comparator): patients received bioactive bonding as lining material then restored with resin composite
  Interventions: Other: patients received bioactive bonding with glass ionomer restorative material

INTERVENTIONS:
Other: patients received calcium hydroxide with glass ionomer restorative material — patients received calcium hydroxide with glass ionomer restorative material
  Arms: patients received calcium hydroxide with resin composite
Other: patients received TheraCal LC with glass ionomer restorative material — patients received TheraCal LC with glass ionomer restorative material
  Arms: patients received TheraCal LC with resin composite
Other: patients received bioactive bonding with glass ionomer restorative material — patients received bioactive bonding with glass ionomer restorative material
  Arms: patients received bioactive bonding with resin composite
Other: patients received universal bonding with glass ionomer restorative material — patients received bioactive bonding with glass ionomer restorative material
  Arms: patients received universal bonding with resin composite

SUMMARY:
The protection of the dentin-pulp complex consists of the application of one or more layers of specific material between the restorative material and dental tissue to avoid additional challenge to the pulp tissue caused by operative procedures, toxicity of restorative materials and bacteria penetration due to microleakage. Protection of the dentinpulp complex has also the function to recover pulp vitality.The materials that can be used for this purpose are varnishes,calcium hydroxide (CH)-based products, glass ionomer cements (GICs) and adhesive systems.The biological compatibility together with the sealing capabilities of dental materials is of paramount importance to avoid or limit pulp tissue irritation and dentinal hypersensitivity.

DETAILED DESCRIPTION:
Pulp plays an important role in the formation and nutrition of dentin as well as in the innervation and defense of the teeth. The primary pulp function is dentin formation, which begins in the moment that the peripheric mesenchimal cells differentiate into odontoblasts and starts the deposition of collagen matrix, in a sequence of deposition/mineralization that ends with the complete tooth formation. Even after the initial formation, pulp continues to physiologically produce dentin due to the tooth aging. Reparative dentin may also be produced in response to physical and/or chemical injuries. Odontoblasts maintain their processes inside the newly formed tissue, thus creating real channels that are responsible for dentin nutrition. changes in the flow of the fluid in the dentinal tubules can trigger pain receptors present on nerve endings in the pulpal aspect to fire nerve impulses, thereby causing pain . This hydrodynamic flow can be increased by changes in temperature, humidity, air pressure and osmotic pressure, or forces acting on the tooth. Hot or cold foods and drinks, and physical pressure are typical triggers in people with dentin hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age ranges from 20-50 years old with vital first permanent molar tooth on testing by vitality test, such as thermal or electrical pulp tester.
2. Class I or II cavities.
3. Deep carious lesions.
4. Absence of clinical signs or symptoms suggesting non-vital tooth such as spontaneous pain, tenderness to percussion, abscess, fistula, periodontal tissue swelling, or abnormal tooth mobility.
5. Sufficient tooth structure for restoration.
6. Healthy patients with good general health.
7. Patients are cooperative and motivated.

Exclusion Criteria:

1. Patient with systemic diseases such as uncontrolled diabetic, cardiovascular diseases, or patient received chemotherapy or radiotherapy.
2. History of spontaneous, unprovoked toothache or mobility, (grade I, II and III).
3. Sensitivity to percussion, external or internal root resorption, periapical lesions or presence of a fistulae.
4. Pregnant females.
5. Drug abuser patients.
6. Previously restored teeth.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Post operative hypersensitivity | 6 month
  Quantitative Assessment by using Verbal analogue scale scoring from 0 - 4 where 0 indicates no pain and 4 indicates intensifying pain

SECONDARY OUTCOMES:
Radiographic evaluation | 6 month
  Patients in all the eight groups were evaluated clinically and radiographically immediately after the procedure,1 week,1 month , 3 months and 6 months using the following criteria: (1) absence of spontaneous pain and/or sensitivity to pressure; (2) absence of sinus, fistula, edema, and/or abnormal mobility; (3) absence of radiolucency at the interradicular and/or periapical regions; (4) absence of internal or external root resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelaziz, PhD, Principal Investigator — BADR University in Cairo
Locations (1):
- Badr University in Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No